CLINICAL TRIAL: NCT05177458
Title: The Effects of Acute Aerobic Exercise on Therapeutic Safety Learning
Brief Title: Exercise and Therapeutic Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Adams (Other)
Responsible Party: Sponsor-Investigator, Thomas Adams, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67199
Record Dates: First submitted 2021-08-12; First posted 2022-01-04 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: PTSD
Keywords: Trauma; Exercise; Mental Health; Aerobic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Exercise (Experimental): Visit 1: Participants will complete study screening, PTSD assessments, and provide written narrative for a traumatic event and a neutral control event.
  Visit 2: Participants will complete eight trials of imaginal exposure (blocks of four neutral and four trauma narrative trials presented as text and sound) with heart rate monitoring and skin conductance. Anxiety will be measured at baseline and after each imagery trial. Participants will then complete 30 minutes of moderate intensity (70-75% maximum heart rate) exercise on a treadmill.
  Visit 3: Participants will complete eight more imaginal trials with heart rate and anxiety ratings as per visit 2.
  Interventions: Behavioral: Experimental
- Control - Low Intensity Exercise (Active Comparator): Visit 1: Participants will complete study screening, PTSD assessments, and provide written narrative for a traumatic event and a neutral control event.
  Visit 2: Participants will complete eight trials of imaginal exposure (blocks of four neutral and four trauma narrative trials presented as text and sound) with heart rate monitoring and skin conductance. Anxiety will be measured at baseline and after each imagery trial. Participants will then complete 30 minutes of light intensity (40-50% maximum heart rate) exercise on a treadmill.
  Visit 3: Participants will complete eight more imaginal trials with heart rate and anxiety ratings as per visit 2.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Experimental — Behavioral: Moderate Intensity Exercise The moderate-intensity aerobic exercise session will consist of walking or running at a moderate intensity (i.e., between 70-75% maximum heart rate) for 30 minutes on a treadmill.
  Arms: Moderate Intensity Exercise
Behavioral: Active Control — Behavioral: Low Intensity Exercise Control participants will maintain light-intensity activity (i.e., walking at 40-50% of maximum heart rate) for 30 minutes.
  Arms: Control - Low Intensity Exercise

SUMMARY:
The proposed project seeks to demonstrate that a brief bout of aerobic exercise can improve a particular type of therapeutic learning among victimins of interpersonal violence with or without posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
The proposed study has one aim:

Specific Aim: To examine the effects of acute exercise on the consolidation of therapeutic safety learning. It is hypothesized that participants who engage in 30-min of moderate-intensity aerobic exercise following the first session of imaginal exposure will show larger between-session (visit 2 to 3) reductions in heart rate and anxiety during imaginal exposure to trauma narratives compared to participants who engage in light-intensity exercise.

ELIGIBILITY:
Inclusion Criteria:

* Experience of interpersonal violence
* English speaking
* Medically healthy

Exclusion Criteria:

* Any endorsed medical concerns related to physical activity (as probed in the phone screening questions regarding cardiovascular, pulmonary, or metabolic disease and as assessed via the Physical Activity Readiness Questionnaire (PAR-Q), which probes into participants' history of heart conditions, chest pain, dizziness, loss of consciousness, bone/joint problems, and medication history). Participants would not be excluded if they report this condition being "controlled" or "addressed" through medication or lifestyle change, such as regular exercise.
* Major medical disorders (such as cancer, AIDS)
* Psychotic disorders
* Intellectual disabilities
* Developmental disorders
* Active substance use disorders
* Pregnancy or probably pregnancy
* Body mass index greater than or equal to 35
* Daily cannabis use
* History of any cardiac disease
* Inability to provide informed consent
* Physical disabilities that prohibit task performance (such as deafness or blindness)
* Self-reported history of loss of consciousness (greater than 30 minutes)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change in participant heart rate | 24 hours (visit 2), 48 hours (visit 3)
  Participant heart rate will be measured at baseline and after each imagery trial using a BIOPAC Bionomadix photo plethysmogram.
Change in participant subjective emotional ratings | 24 hours (visit 2), 48 hours (visit 3)
  Participant anxiety will be measured at baseline and after each imagery trial.
Change in participant electrodermal response | 24 hours (visit 2), 48 hours (visit 3)
  Participant skin conductance activity will be measured at baseline and during each imagery trial using a pair of BIOPAC Bionomadix electrodermal activity electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Adams Jr, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No